CLINICAL TRIAL: NCT02847507
Title: Seroprevalence of Hepatitis E in HIV Positive Patients in Basque Country in 2016 (VIhVhEpb): a Prospective Cohort Study
Brief Title: Seroprevalence of Hepatitis E in HIV Positive Patients in Basque Country in 2016 (VIhVhEpb)
Acronym: VIhVhEpb
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de la côte Basque (Other)
Collaborators: University Hospital, Toulouse (Other)
Responsible Party: Principal Investigator, VAREIL Marc-Olivier, doctor, Centre Hospitalier de la côte Basque
Other Study IDs: VIH VHE pays basque
Record Dates: First submitted 2016-07-20; First posted 2016-07-28 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: HIV; Hepatitis E
Keywords: HIV; Hepatitis E
MeSH Terms: conditions — Hepatitis E

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serological status for hepatitis E, hepatits B and hepatitis C, and biological follow up of HIV patients including fibrotest for hepatis b/ or C positive patients
Oversight: Data Monitoring Committee: No

SUMMARY:
Study of seroprevalence of hepatitis E among HIV positive patient in Basque country, France in 2016.

DETAILED DESCRIPTION:
Study of seroprevalence of hepatitis E among patient followed and treated in "centre Hospitalier de la Côte Basque" for HIV infections. Study of acquisition of hepatitis E , and determination of liver status using fibrotest in co-infected patients with hepatis C and / or B.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive > 18

Exclusion Criteria:

* patient refusal for participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients seropositve for HIV and treated in the" Centre Hospitalier de la côte Basque" are considered for enrollment.
  Patient must be > 18 years, and followed or treated in the investigators institution
Sampling Method: Non-Probability Sample
Enrollment: 307 (Actual)
Dates: Start 2016-07; Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of immunoglobulin M (IgM) and Immunoglobulin G (IgG) for hepatitis E in blood sample of each patients. Positive sample for both IgM and IgG will be confirmed using polymerase chain reaction (PCR) techniques | 6 months time period
  Blood samples will be tested for specific immunoglobulins against hepatitis E virus

SECONDARY OUTCOMES:
fibrotest score | 6 months time period
  patients infected with hepatitis B or hepatitis C viruses will have their liver status determined using fibrotest score.

CONTACTS AND LOCATIONS:
Overall Officials: Marc-olivier Vareil, phd, Principal Investigator — centre hospitalier côte Basque
Locations (1):
- Centre hospitalier de la Côte Basque, Bayonne, France

IPD SHARING:
Plan to Share IPD: Undecided